CLINICAL TRIAL: NCT01094327
Title: Evaluation of Recipients With and Without Proteinuria, Pre and Post Kidney Transplantation
Brief Title: Proteinuria in Pre and Post Transplant
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, George W. Burke, Professor of Surgery, University of Miami
Other Study IDs: 20070206
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Proteinuria
Keywords: focal segmental glomerulosclerosis
MeSH Terms: conditions — Proteinuria; Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with focal segmental glomerulosclerosis (FSGS) who progress rapidly to end stage renal disease (ESRD) are at highest risk for development of recurrence of proteinuria following kidney transplantation. This study will look at serum specimens pre and post transplant, as well as kidney transplant specimens pre and post reperfusion to identify where the defects has occured that results in recurrence of proteinuria in a given kidney transplant.

DETAILED DESCRIPTION:
This study will retrospectively review patient's medical records for protein in the urine, blood creatinine and kidney biopsy results. Also character of the fluid used to flush the kidney before transplant will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients
* Pediatric males and females up to the age of 25 years old.

Exclusion Criteria:

* Transplant recipients other than kidney

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric population up to the age of 25 years old, with biopsy diagnosed of FSGS (focal segmental glomerulosclerosis).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-02 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Explain mechanisms behind the development of proteinuria in patients immediately after receiving a kidney transplant | through study completion, an average of 5 years
  chart review

CONTACTS AND LOCATIONS:
Overall Officials: George Burke, M.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine Transplant Clinic, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No